CLINICAL TRIAL: NCT06405633
Title: A Phase 1b/2a Open-label Single Ascending Doses (SAD) and Multiple Ascending Doses (MAD) Research Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Participants With AATD Pi*ZZ on WVE-006 (RestorAATion-2)
Brief Title: A Phase 1b/2a, Open-label Single Ascending Doses and Multiple Ascending Doses Study in Participants With Pi*ZZ AATD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WVE-006-002
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- WVE-006 (Dose 1) (Experimental)
  Interventions: Drug: WVE-006
- WVE-006 (Dose 2) (Experimental)
  Interventions: Drug: WVE-006
- WVE-006 (Dose 3) (Experimental)
  Interventions: Drug: WVE-006

INTERVENTIONS:
Drug: WVE-006 — RNA editing oligonucleotide

SUMMARY:
The purpose of this open-label study is to assess the safety, tolerability, pharmacodynamics, and pharmacokinetics of WVE-006 in participants with alpha-1 antitrypsin deficiency (AATD) following Period 1 single ascending dose (SAD) and Period 2 multiple ascending doses (MAD), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the Investigator, based on a medical evaluation, or has mild to moderate AATD-induced lung disease (FEV1 ≥50%) and/or stable mild AATD-induced liver disease (≤F2 (≤10 kPa) on FibroScan.
* Genetic testing confirming Pi*ZZ.
* Participant has been a non-smoker for at least 1 year prior to screening.

Exclusion Criteria:

* • Participant has a history of multiple drug allergies or of allergic reaction to an oligonucleotide or to N-acetylgalactosamine (GalNAc).

  * Participant has a history of intolerance or any medical condition that might interfere with subcutaneous injections.
  * Any ongoing or recent infections.
  * Any recent or planned vaccinations during the study.
  * Participant has a history of regular alcohol consumption exceeding 14 standard drinks/week.
  * Unwilling to abstain from alcohol for 48 hours prior to dosing at each of the dosing visits.
  * Any recent or planned major surgery during the study.
  * Participant has any medical condition or social circumstance that, in the opinion of the Investigator, would make the participant unsuitable for participation in the study or for dosing on Day 1, or could interfere with the assessments of safety, pharmacodynamics, or pharmacokinetics, or completion of the study.
  * Participant currently on AAT augmentation therapy, planned to be on augmentation therapy anytime during the study, or has been on augmentation therapy within 30 days prior to Screening Visit.
  * Donation of blood or blood products in excess of 500 mL within 12 weeks prior to Screening Visit and/or unwilling to refrain from blood donation for the duration of the study.
  * Participant has received an investigational agent within 3 months of the Screening Visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with adverse events | Up to 36 Weeks

SECONDARY OUTCOMES:
Single Ascending Dose - Change from baseline in levels of serum M-AAT protein. | Up to 12 Weeks
Multiple Ascending Dose - Change from baseline in levels of serum M-AAT protein | Up to 24 Weeks
Single Ascending Dose - Area under the plasma concentration time curve for WVE-006 from time of dosing to the last measurable concentration (AUClast) | Up to 12 Weeks
Single Ascending Dose - Maximum concentration of WVE-006 in plasma | Up to 12 Weeks
Multiple Ascending Doses - Area under the plasma concentration time curve for WVE-006 from time of dosing to the last measurable concentration (AUClast) | Up to 24 Weeks
Multiple Ascending Doses - Maximum concentration of WVE-006 in plasma (Cmax) | Up to 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Caracta, MD, Study Director — Wave Life Sciences
Locations (9):
- St. Vincent's Hospital, Melbourne, Fitzroy, Victoria, Australia
- Canada (2):
  - Dalhousie University - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Inspiration Research Limited, Toronto, Ontario
- Turku University Hospital, Turku, Finland
- Universitaetsklinikum Aachen, AoeR, Aachen, Germany
- Waikato Hospital, Hamilton, New Zealand
- United Kingdom (3):
  - Queen Elizabeth Hospital, University Hospital Birmingham, Birmingham
  - Cambridge University - Addenbrooke's Hospital, Cambridge
  - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No